CLINICAL TRIAL: NCT04759287
Title: Effectiveness of C-MAC Video-stylet Versus Fiberoptic Bronchoscope for Awake Intubation in Patients With Predicted Difficult Airway
Brief Title: Effectiveness of C-MAC Video-stylet Versus Fiberoptic Bronchoscope for Awake Intubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: rehab zayed (Other)
Responsible Party: Sponsor-Investigator, rehab zayed, Assisstant Professor of Anesthesia, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 0304792
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Difficult Mask Ventilation; Difficult Intubation

STUDY DESIGN:
Intervention Model Description: The patients will be randomly assigned into two equal groups using computer-generated randomization technique. The first group (VS group) will include patients undergoing awake intubation using the C-MAC VS. The second control group (FOB group) will include patients undergoing awake intubation using the flexible fibreoptic bronchoscope.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VS group (Active Comparator): include patients undergoing awake intubation using the C-MAC VS
  Interventions: Device: C-MAC VS
- FOB group (Placebo Comparator): will include patients undergoing awake intubation using the flexible fibreoptic bronchoscope.
  Interventions: Device: flexible fibreoptic bronchoscope

INTERVENTIONS:
Device: C-MAC VS — The first group (VS group) will include patients undergoing awake intubation using the C-MAC VS
  Arms: VS group
Device: flexible fibreoptic bronchoscope — The second control group (FOB group) will include patients undergoing awake intubation using the flexible fibreoptic bronchoscope.
  Arms: FOB group

SUMMARY:
C-MAC- Video Stylet is a completely new type of video endoscope. It combines the advantages of both rigid and flexible intubation endoscopes.

DETAILED DESCRIPTION:
C-MAC-VS can be connected easily to the same C- MAC monitor and Pocket Monitor without requiring any additional light source and camera. This device is great for cases with limited mouth opening, airway obstruction and difficult intubation.

ELIGIBILITY:
Inclusion Criteria:

* patients with BMI ≥ 30 kg/m2,
* presence of any predictors of difficult intubation;
* Mallampati score > =3;
* inter-incisor distance < 3 cm;
* thyromental distance < 6 cm;
* neck extension < 80°from neck flexion;
* cervical spine instability;
* history of difficult endotracheal intubation or difficult mask ventilation

Exclusion Criteria:

* patients have increased risk of pulmonary aspiration;
* have significant medical diseases in term of cardiac, respiratory, hepatic, renal,

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-05-20 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
the time required for a wake intubation | 10 minutes
  assess the time required for a wake intubation using C-MAC VS versus FOB in patients with anticipated difficult airway.

CONTACTS AND LOCATIONS:
Overall Officials: rehab A. Abd Elaziz, Ass.Prof., Principal Investigator — Alexandria University
Locations (1):
- rehab Abd Elaziz, Alexandria, Egypt